CLINICAL TRIAL: NCT02294903
Title: A Prospective Development Study Evaluating Focal Therapy Using Encage Coiled Bipolar Radiofrequency Ablation in Men With Localised Prostate Cancer
Brief Title: Focal Prostate Radiofrequency Ablation
Acronym: ProRAFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trod Medical N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TM-105
Record Dates: First submitted 2014-11-15; First posted 2014-11-19 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Prostate Cancer
Keywords: Focal radiofrequency ablation; Prostate cancer; Encage
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ProRAFT (Experimental): Procedure/Surgery: Coiled Bipolar Radiofrequency Ablation
  Interventions: Procedure: Coiled Bipolar Radiofrequency Ablation

INTERVENTIONS:
Procedure: Coiled Bipolar Radiofrequency Ablation — Radiofrequency ablation by use of bipolar electrodes

SUMMARY:
To assess the early histological outcomes of tissue ablation, adverse events and genitourinary side-effect profile of focal radiofrequency ablation using a coiled bipolar device to treat localized prostate cancer in men with clinically significant prostate cancer.

DETAILED DESCRIPTION:
The study aims to assess the ability of focal therapy using coiled bipolar radiofrequency device to ablate a pre-defined target tissue zone as well as assess side-effects. The medical device has a coiled configuration and creates thus a "Faraday cage" effect, preventing surrounding tissue damage and the bipolar configuration produces complete tissue thermo coagulation within the limits the coil.

Thereof it is proposed to conduct a prospective development study, offering focal therapy coiled bipolar radiofrequency ablation to men with histologically proven localized prostate cancer which is clinically significant.

Localization and characterization of the disease will be established using multi-parametric magnetic resonance imaging (mp-MRI) and transperineal prostate biopsies. Magnetic resonance (MR)-visible, clinically significant disease will be targeted and focally treated with a margin of normal tissue as big as anatomically possible to obtain an adequate margin of normal tissue around the lesion for effective ablation. Secondary lesions meeting criteria for clinical insignificance will be left untreated and undergo surveillance.

Pre-operative and all post operative imaging will be performed using a scanner and a pelvic phased array receiver, with a pelvic coil. A full protocol of T1 and T2 weighted turbo-spin echo images and a dynamic post gadolinium volume acquisition will be used for both pre-operative diagnostic and planning scans and post-operative assessment by use of the medical device.

The initial transperineal biopsy will already have been performed, prior to invitation to participate in the study, and demonstrating eligibility for inclusion.

The process will involve targeted or mapping biopsies which are concordant with the lesion seen on MRI. In both cases, transperineal biopsies will be taken from the prostate using a brachytherapy grid placed over the perineal skin whilst the man is in the lithotomy position.

They will be given as much time as they need to consider whether or not patients wish to participate. The ones who wish to participate after reading the patient information sheet will undergo a screening visit (first visit) to ascertain whether or not they are eligible for the trial. If so, they will proceed to focal radiofrequency ablation using a coiled bipolar device(second visit), and will be seen at further follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate cancer
* A visible lesion on multiparametric Magnetic Resonance Imaging (mpMRI), that is accessible to a treatment based on radiofrequency bipolar electrodes
* Transperineal prostate biopsies (template mapping and/or targeted) correlating with clinically significant lesion in the area of the Magnetic Resonance (MR)-visible lesion
* Absence of clinically significant histological disease outside of the planned treatment zone
* Radiological stage T1-T3aN0M0 disease, as determined by local guidelines
* Serum prostate-specific antigen (serum PSA) </=15ng/ml within 3 months of screening visit
* Life expectancy of more than 10 years
* Signed informed consent by patient
* An understanding of the English language sufficient to understand written and verbal information about the trial and consent process

Exclusion Criteria:

* Men who have had previous radiation therapy to the pelvis
* Men who have had androgen suppression/hormone treatment within the previous 12 months for their prostate cancer
* Men with evidence of metastatic disease or nodal disease outside the prostate on bone scan or cross-sectional imaging
* Men with a tumour not visible on mpMRI
* Men with an inability to tolerate a transrectal ultrasound (TRUS)
* Men allergic to latex
* Men who have undergone prior significant rectal surgery preventing insertion of the transrectal ultrasound probe (decided on the type of surgery in individual cases)
* Men who have had previous electroporation, radiofrequency ablation, High Intensity Focused Ultrasound (HIFU), cryosurgery, thermal or microwave therapy to the prostate
* Men who have undergone a Transurethral Resection of the Prostate (TURP) for symptomatic lower urinary tract symptoms within the prior 6 months. These patients may be included within the trial if deferred from consent and screening until at least 6 months following the TURP
* Men not fit for major surgery as assessed by a Consultant Anaesthetist
* Men unable to have pelvic MRI scanning (severe claustrophobia, permanent cardiac pacemaker, metallic implant etc likely to contribute significant artefact to images)
* Presence of metal implants/stents in the urethra
* Men with renal impairment with a Glomerular Filtration Rate (GFR) of <35ml/min (unable to tolerate Gadolinium dynamic contrast enhanced MRI)

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
Cancer control outcome | 6 months
  To determine the ablative efficacy of focal therapy to treat localized low to intermediate risk prostate cancer using coiled bipolar radiofrequency ablation (Encage)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed U HASHIM, FRCS, PhD, Study Chair — UCLH NHS Foundation Trust; Mark EMBERTON, FRCS, MD, Principal Investigator — Division of Surgery & Interventional Science, UCL
Locations (1):
- University College London Hospitals, London, United Kingdom